CLINICAL TRIAL: NCT00498303
Title: A Phase III, Multicenter, Uncontrolled, Open-Label Study to Evaluate Safety and Immunogenicity of Preservative Free, Inactivated Split Influenza Vaccine, Using the Strain Composition 2007/2008 When Administered to Adult and Elderly Subjects
Brief Title: Safety and Immunogenicity of Trivalent Split Influenza Vaccine Using the Strain Composition 2007/2008
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V44P11S; 2007-001403-38
Record Dates: First submitted 2007-07-09; First posted 2007-07-10 (Estimated); Last update posted 2008-04-22 (Estimated); Status verified 2008-04

CONDITIONS: Seasonal Influenza; Vaccine
Keywords: influenza vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: trivalent split influenza vaccine

SUMMARY:
Annual trial for registration of trivalent split influenza vaccine with the strain composition of the season 2007/2008 in healthy adult and elderly subjects

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age, mentally competent, willing and able to give informed consent prior to study entry
* available for all the visits scheduled in the study and able to comply with all study requirements
* in good health as determined by: medical history, physical examination, clinical judgment of the investigator

Exclusion Criteria:

* n/a

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2007-06

PRIMARY OUTCOMES:
evaluate the antibody response to each influenza vaccine antigen, as measured by haemagglutination inhibition (HI) test on Day 0 and on Day 21
evaluate safety of trivalent split influenza vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (1):
- Werksarztzentrum Herborn, Herborn, Germany